CLINICAL TRIAL: NCT00477269
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of the Six Months Treatment With the Tyrosine Kinase Inhibitor STI571 for the Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: Safety and Efficacy of Imatinib Mesylate in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSTI571E2203; 2005-005569-12
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension, tyrosine kinase inhibitor, STI571
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- STI571 (Experimental): STI571
  Interventions: Drug: Imatinib mesylate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- All Patients (Experimental): Open label extension
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate
  Other Names: Imatinib, Glivec, Gleevec, STI571, QTI571
  Arms: All Patients; STI571
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of imatinib mesylate in patients with pulmonary arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAH of either primary (idiopathic), familial or secondary to systemic sclerosis (excluding those with marked pulmonary fibrosis) according to World Conference on Pulmonary Hypertension classification (Venice, 2003).
* Symptoms with a WHO class of II-IV

Exclusion Criteria:

* Use of unspecific phosphodiesterase inhibitors (for example, pentoxyfillin, enoximon, milrinone or pimobendan) during the study
* Chronic inhaled nitric oxide therapy from start to study completion
* Treatment with catecholamines (for example, adrenalin, noradrenalin, dopamine),
* Pre-existing lung diseases, including parasitic diseases affecting lungs, asthma, congenital abnormalities of the lungs, chest, and diaphragm.
* Pulmonary artery or valve stenosis; pulmonary venous hypertension; chronic thromboembolic pulmonary hypertension
* Acute heart failure or chronic left sided heart failure; congenital or acquired valvular or myocardial disease
* Severe (systemic) arterial hypertension (> 200 mmHg (systolic) or > 120 mmHg (diastolic)) Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis, Principal Investigator — Investigative site
Locations (13):
- United States (3):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis investigative site, Newark, New Jersey
  - Novartis Investigative Site, New York, New York
- Austria (2):
  - Novartis Investigative Site, Graz, Austria
  - Novartis Investigative site, Graz
- Germany (4):
  - Novartis Investigative Site, Hanover, Germany
  - Novartis Investigative Site, Giessen
  - Novartis Investigative site, Giessen
  - Novartis Investigative site, Hanover
- United Kingdom (4):
  - Novartis Investigative Site, Cambridge, Cambridgeshire
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative site, Glasgow
  - Novartis Investigative site, Papworth Everard

REFERENCES:
- [Derived] Ghofrani HA, Morrell NW, Hoeper MM, Olschewski H, Peacock AJ, Barst RJ, Shapiro S, Golpon H, Toshner M, Grimminger F, Pascoe S. Imatinib in pulmonary arterial hypertension patients with inadequate response to established therapy. Am J Respir Crit Care Med. 2010 Nov 1;182(9):1171-7. doi: 10.1164/rccm.201001-0123OC. Epub 2010 Jun 25. PMID 20581169

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 42 participants that completed the Core Study only 22 Participants continued into the Open Label Extension. Not all participants were required to continue into the extension from the core.
Period: Core Study
Arm/Group | STI571 | Placebo | All Patients
Started | 28 | 31 | 0
Completed | 19 | 23 | 0
Not Completed | 9 | 8 | 0
Not completed — Adverse Event | 6 | 4 | 0
Not completed — Death | 3 | 3 | 0
Not completed — Withdrawn Consent | 0 | 1 | 0
Period: Open Label Extension
Arm/Group | STI571 | Placebo | All Patients
Started | 0 (Arm in the Core study not extension) | 0 (Arm in the Core study not extension) | 22
Completed | 0 (Arm in the Core study not extension) | 0 (Arm in the Core study not extension) | 9
Not Completed | 0 | 0 | 13
Not completed — Adverse Event | 0 | 0 | 4
Not completed — Abnormal laboratory values | 0 | 0 | 1
Not completed — unsatisfactory therapeutic effects | 0 | 0 | 2
Not completed — Adminiatrative problems | 0 | 0 | 2
Not completed — Death | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STI571 | Placebo | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (15.3) | 44.2 (15.7) | 44.3 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 22 | 40
  Male | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs), Serious Adverse Events (SAEs) and Death During the Core
Description: In this analysis patients with all (serious and non -serious) adverse events, and death were reported. See Safety Section.
Time Frame: 6 months
Population: Safety Population all participants enrolled was included in this population
Measure: Number; unit: participants
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
participants
  Paients with AE(s) | 27 | 29
  Death | 3 | 3
  SAE(s) | 12 | 11

2. Primary Outcome: Number of Patients With Adverse Events (AEs), Serious Adverse Events (SAEs) and Death During the Extension
Description: as for outcome 1
Time Frame: 72 months
Population: No formal statistical analysis was performed in the extension phase of this study so no analysis data sets were defined. All summaries are based on all patients enrolled.
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 22
participants
  Any AE(s) | 22
  Death | 4
  SAE(s) | 16

3. Primary Outcome: Change From Baseline of Six Minute Walk Test - Total Distance Walked at Different Time Periods
Description: The Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Distance <500 meters suggests considerable exercise limitation; Distance 500-800 meters suggests moderate limitation; Distance >800 meters (with no rests) suggests mild or no limitation.
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
meters
  Day 32 (n=25,27) | 10.2 (53.7) | 8.2 (27.5)
  week 8 (n=23,24) | 17.0 (55.6) | 15.5 (40.8)
  week 12 (n=22,24) | 21 (36.2) | 7.8 (50.0)
  week 16 (n=19, 23) | 25.5 (43.1) | 12.1 (47.9)
  week 20 (n=19, 21) | 38.3 (42.5) | 12.8 (60.4)
  study completion Week 24 (n=21, 12) | 22.0 (63.1) | -1.0 (53.3)

4. Primary Outcome: Change From Baseline of Six Minute Walk Test - Number of Stops at Different Time Periods
Description: The Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Number of stops were recorded for each patient.
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: number of stops
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
number of stops
  Day 32 (n=25,27) | -0.2 (0.7) | 0.1 (0.4)
  week 8 (n=23,24) | -0.2 (0.7) | 0.0 (1.1)
  week 12 (n=22,24) | -0.3 (0.9) | 0.3 (0.9)
  week 16 (n=19, 23) | -0.3 (0.8) | 0.0 (0.2)
  week 20 (n=19, 21) | -0.4 (1.0) | 0.3 (1.0)
  study completion Week 24 (n=21, 12) | -0.3 (0.8) | -0.1 (0.5)

5. Primary Outcome: Change From Baseline of Six Minute Walk Test - Total Duration of Stops at Different Time Periods
Description: The Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. If the patient stopped the duration of each stop was recorded.
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
minutes
  Day 32 (n=25,27) | -0.06 (0.19) | 0.12 (0.36)
  week 8 (n=23,24) | -0.03 (0.10) | 0.07 (0.27)
  week 12 (n=22,24) | -0.03 (0.10) | 0.19 (0.55)
  week 16 (n=19, 23) | -0.03 (0.10) | 0.06 (0.26)
  week 20 (n=19, 21) | -0.05 (0.15) | 0.12 (0.42)
  study completion Week 24 (n=21, 12) | -0.02 (0.10) | 0.03 (0.18)

6. Secondary Outcome: Number of Patients With Pulmonary Hypertension (PAH) Assessd by World Health Organization (WHO) Classification on Physical Activity
Description: PAH assessed according to the WHO classification: Class I Patients with PAH but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near syncope. Class II Patients with PAH resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope. Class III Patients with PAH resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes undue dyspnea or fatigue, chest pain or near syncope. Class IV Patients with PAH with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may even be present at rest. Discomfort is increased by any physical activity.
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Number; unit: number of participants
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
number of participants
  Baseline: WHO Class IV (n=27,30) | 2 | 1
  Baseline: WHO Class III (n=27,30) | 14 | 22
  Baseline: WHO Class II (n=27,30) | 11 | 7
  Day 32: WHO Class IV (n=27,30) | 3 | 3
  Day 32: WHO Class III (n=27,30) | 11 | 21
  Day 32: WHO Class II (n=27,30) | 13 | 6
  Week 8: WHO Class IV (n=24,27) | 3 | 1
  Week 8: WHO Class III (n=24,27) | 9 | 20
  Week 8: WHO Class II (n=24,27) | 12 | 6
  Week 12: WHO Class IV (n=23,27) | 0 | 1
  Week 12: WHO Class III (n=23,27) | 12 | 17
  Week 12: WHO Class II (n=23,27) | 11 | 9
  Week 16: WHO Class IV (n=22,27) | 0 | 1
  Week 16: WHO Class III (n=22,27) | 11 | 18
  Week 16: WHO Class II (n=22,27) | 11 | 7
  Week 16: WHO Class I (n=22,27) | 0 | 1
  Week 20: WHO Class IV (n=19,24) | 0 | 1
  Week 20: WHO Class III (n=19,24) | 10 | 14
  Week 20: WHO Class II (n=19,24) | 8 | 9
  Week 20: WHO Class I (n=19,24) | 1 | 0
  Week 24: WHO Class IV (n=21,25) | 1 | 2
  Week 24: WHO Class III (n=21,25) | 12 | 13
  Week 24: WHO Class II (n=21,25) | 8 | 10

7. Secondary Outcome: Borg Score-Oxygen Saturation(SaO2) During the Six Minutes Walk Test at Different Time Periods
Description: Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. During the walk the patient was connected to a portable pulse oximeter via a finger probe. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. The test was terminated if the patient became too distressed or if their SaO2% fell below 60%.
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Percentage of Oxygen Saturation
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
Percentage of Oxygen Saturation
  Baseline: Resting (n= 28, 29) | 94.3 (4.6) | 93.4 (4.7)
  Baseline: End of Test (n= 28, 28) | 87.9 (12.4) | 87.9 (8.2)
  Baseline: 2 minutes after end of test (n=26, 26) | 93.0 (7.0) | 92.0 (6.2)
  Day 32: Resting (n= 25, 28) | 94.5 (4.0) | 92.4 (6.3)
  Day 32: End of Test (n= 25, 28) | 89.0 (11.2) | 87.2 (12.8)
  Day 32: 2 minutes after end of test (n= 25, 26) | 94.8 (4.6) | 92.7 (7.1)
  Week 8: Resting (n= 23, 25) | 95.1 (3.3) | 93.2 (6.1)
  Week 8: End of Test (n= 23, 24) | 90.9 (6.7) | 87.9 (11.9)
  Week 8: 2 minutes after end of test (n= 23, 23) | 94.4 (5.3) | 93.1 (7.8)
  Week 12: Resting (n= 22, 25) | 95.1 (4.8) | 93.9 (5.6)
  Week 12: End of Test (n= 20, 24) | 89.8 (9.2) | 89.6 (8.9)
  Week 12: 2 minutes after end of test (n= 19, 22) | 92.7 (8.9) | 94.2 (5.6)
  Week 16: Resting (n= 19, 24) | 95.0 (5.0) | 94.1 (5.1)
  Week 16: End of Test (n= 18, 23) | 87.9 (13.1) | 88.1 (9.8)
  Week 16: 2 minutes after end of test (n= 19, 19) | 94.6 (6.0) | 93.3 (8.0)
  Week 20: Resting (n= 19, 22) | 94.0 (4.7) | 93.7 (5.0)
  Week 20: End of Test (n= 18, 21) | 87.5 (13.2) | 87.6 (9.1)
  Week 20: 2 minutes after end of test (n= 19, 21) | 93.8 (7.1) | 93.4 (7.4)
  Week 24: Resting (n= 20, 22) | 95.5 (3.4) | 94.3 (4.6)
  Week 24: End of Test (n= 20, 21) | 89.9 (7.1) | 89.3 (8.4)
  Week 24: 2 minutes after end of test (n= 20, 21) | 94.8 (4.3) | 94.8 (3.9)

8. Secondary Outcome: Borg Score-Systolic Blood Pressure During the Six Minutes Walk Test at Different Time Periods
Description: Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. During the walk the patient was connected to a portable pulse oximeter via a finger probe. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Systolic blood pressure (mmHg) were recorded before the test at resting, at the end of the test and two minutes after the end of the test
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline: Resting (n= 26, 28) | 111.3 (14.2) | 104.6 (13.2)
  Baseline: End of Test (n= 21, 26) | 119.9 (19.3) | 118.3 (18.0)
  Baseline: 2 minutes after end of test (n=25, 27) | 120.0 (18.3) | 110.4 (13.6)
  Day 32: Resting (n= 25, 27) | 111.4 (9.6) | 106.0 (12.3)
  Day 32: End of Test (n= 22, 22) | 126.5 (17.3) | 122.3 (18.6)
  Day 32: 2 minutes after end of test (n= 25, 26) | 119.6 (12.6) | 113.8 (14.9)
  Week 8: Resting (n= 22, 24) | 108.9 (12.3) | 107.3 (13.5)
  Week 8: End of Test (n= 19, 20) | 124.6 (16.1) | 119.9 (17.1)
  Week 8: 2 minutes after end of test (n= 23, 24) | 115.2 (13.6) | 114.5 (13.7)
  Week 12: Resting (n= 22, 23) | 106.5 (11.5) | 107.7 (13.8)
  Week 12: End of Test (n= 17, 19) | 122.2 (17.0) | 118.8 (22.9)
  Week 12: 2 minutes after end of test (n= 20, 22) | 115.9 (14.2) | 115.9 (14.9)
  Week 16: Resting (n= 19, 22) | 106.7 (9.7) | 105.7 (12.5)
  Week 16: End of Test (n= 15,18) | 117.2 (12.3) | 119.8 (13.5)
  Week 16: 2 minutes after end of test (n= 19, 22) | 114.6 (13.8) | 112.6 (15.8)
  Week 20: Resting (n= 19, 20) | 106.5 (7.0) | 109.1 (12.1)
  Week 20: End of Test (n= 16,17) | 122.4 (13.3) | 119.9 (19.3)
  Week 20: 2 minutes after end of test (n= 19, 20) | 115.5 (14.0) | 115.1 (15.1)
  Week 24: Resting (n= 20, 21) | 110.6 (15.6) | 108.2 (15.7)
  Week 24: End of Test (n= 16, 17) | 126.9 (23.6) | 116.8 (14.9)
  Week 24: 2 minutes after end of test (n= 20, 19) | 118.2 (18.6) | 111.1 (10.6)

9. Secondary Outcome: Borg Score-Diastolic Blood Pressure During the Six Minutes Walk Test at Different Time Periods
Description: Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. During the walk the patient was connected to a portable pulse oximeter via a finger probe. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Diastolic blood pressure (mmHg) were recorded before the test at resting, at the end of the test and two minutes after the end of the test
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline: Resting (n= 26, 28) | 68.2 (10.2) | 67.9 (8.9)
  Baseline: End of Test (n= 21, 26) | 75.1 (10.8) | 69.5 (11.9)
  Baseline: 2 minutes after end of test (n=25, 27) | 71.6 (9.8) | 67.9 (9.6)
  Day 32: Resting (n= 25, 27) | 69.6 (10.4) | 68.4 (8.8)
  Day 32: End of Test (n= 22, 22) | 78.2 (12.3) | 75.2 (11.2)
  Day 32: 2 minutes after end of test (n= 25, 26) | 72.5 (9.1) | 70.7 (9.4)
  Week 8: Resting (n= 22, 24) | 67.7 (11.8) | 68.8 (9.0)
  Week 8: End of Test (n= 19, 20) | 74.8 (10.8) | 74.0 (10.9)
  Week 8: 2 minutes after end of test (n= 23, 24) | 71.2 (10.3) | 72.2 (11.7)
  Week 12: Resting (n= 22, 23) | 65.5 (8.3) | 70.6 (11.6)
  Week 12: End of Test (n= 17, 19) | 75.6 (11.5) | 72.4 (14.3)
  Week 12: 2 minutes after end of test (n= 20, 22) | 73.1 (8.9) | 72.0 (13.7)
  Week 16: Resting (n= 19, 22) | 67.7 (9.9) | 66.7 (7.7)
  Week 16: End of Test (n= 15,18) | 72.7 (9.2) | 76.7 (8.6)
  Week 16: 2 minutes after end of test (n= 19, 22) | 71.4 (11.0) | 70.5 (8.0)
  Week 20: Resting (n= 19, 20) | 67.2 (8.0) | 69.8 (8.8)
  Week 20: End of Test (n= 16,17) | 72.9 (8.7) | 72.9 (8.1)
  Week 20: 2 minutes after end of test (n= 19, 20) | 71.9 (9.2) | 72.7 (9.8)
  Week 24: Resting (n= 20, 21) | 69.7 (10.3) | 70.7 (10.9)
  Week 24: End of Test (n= 16, 17) | 74.1 (10.7) | 72.3 (10.9)
  Week 24: 2 minutes after end of test (n= 20, 19) | 71.3 (10.1) | 72.9 (9.5)

10. Secondary Outcome: Borg Score-Heart Rate (HR) During the Six Minutes Walk Test at Different Time Periods
Description: Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. During the walk the patient was connected to a portable pulse oximeter via a finger probe. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Heart Rate (bpm) were recorded before the test at resting, at the end of the test and two minutes after the end of the test
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
beats per minute (bpm)
  Baseline: Resting (n= 28, 29) | 80.8 (13.0) | 87.9 (12.7)
  Baseline: End of Test (n= 28, 29) | 106.3 (23.9) | 112.3 (20.4)
  Baseline: 2 minutes after end of test (n=26, 26) | 84.2 (16.9) | 94.1 (14.6)
  Day 32: Resting (n= 25, 28) | 80.7 (14.3) | 83.6 (15.7)
  Day 32: End of Test (n= 25, 28) | 108.4 (19.1) | 113.1 (19.5)
  Day 32: 2 minutes after end of test (n= 25, 26) | 89.2 (17.0) | 90.6 (14.1)
  Week 8: Resting (n= 23, 25) | 80.3 (9.6) | 81.1 (11.2)
  Week 8: End of Test (n= 23, 24) | 109.5 (21.4) | 110.3 (26.4)
  Week 8: 2 minutes after end of test (n= 23, 23) | 85.3 (15.7) | 88.9 (13.2)
  Week 12: Resting (n= 22, 25) | 76.5 (13.2) | 85.1 (13.2)
  Week 12: End of Test (n= 20, 25) | 105.3 (26.2) | 113.0 (26.5)
  Week 12: 2 minutes after end of test (n= 19, 22) | 83.8 (17.8) | 89.4 (15.7)
  Week 16: Resting (n= 19, 24) | 76.5 (13.2) | 84.4 (12.9)
  Week 16: End of Test (n= 18, 23) | 102.8 (25.6) | 117.9 (24.3)
  Week 16: 2 minutes after end of test (n= 19, 21) | 85.8 (21.0) | 85.5 (14.4)
  Week 20: Resting (n= 19, 22) | 75.3 (13.8) | 80.2 (9.6)
  Week 20: End of Test (n= 18,22) | 109.2 (26.8) | 118.0 (24.5)
  Week 20: 2 minutes after end of test (n= 19, 21) | 83.3 (17.4) | 87.3 (11.4)
  Week 24: Resting (n= 20, 22) | 79.5 (13.8) | 83.6 (8.6)
  Week 24: End of Test (n= 20, 21) | 110.2 (18.1) | 116.8 (21.7)
  Week 24: 2 minutes after end of test (n= 20, 21) | 87.9 (17.5) | 88.9 (11.8)

11. Secondary Outcome: Borg Score During the Six Minutes Walk Test at Different Time Periods
Description: Borg Score during Six Minute Walk test was carried out along a course, such as a hospital corridor, measuring at least 20 meters delineated by markers. During the walk the patient was connected to a portable pulse oximeter via a finger probe. Patients were instructed to walk at a comfortable speed as far as they could manage in six minutes, resting whenever they needed to. Borg Score of Breathlessness was recorded using the following score of 0 to 10, how breathless do you feel? 0 is nothing at all and 10 is maximal breathlessness
Time Frame: Baseline, Day 32, Week 8, Week 12, Week 16, Week 20 and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
score on a scale
  Baseline: Resting (n= 26, 27) | 0.27 (0.83) | 0.43 (0.92)
  Baseline: End of Test (n= 27, 29) | 3.34 (2.30) | 3.02 (1.59)
  Baseline: 2 minutes after end of test (n=24, 26) | 0.88 (1.67) | 1.08 (1.47)
  Day 32: Resting (n= 25, 27) | 0.24 (0.83) | 0.48 (0.86)
  Day 32: End of Test (n= 25, 28) | 2.53 (2.02) | 3.07 (2.08)
  Day 32: 2 minutes after end of test (n= 25, 26) | 0.65 (2.06) | 1.06 (1.34)
  Week 8: Resting (n= 23, 24) | 0.32 (1.02) | 0.38 (0.81)
  Week 8: End of Test (n= 23, 25) | 2.46 (2.02) | 2.32 (1.64)
  Week 8: 2 minutes after end of test (n= 23, 24) | 0.32 (0.92) | 0.58 (1.04)
  Week 12: Resting (n= 22, 24) | 0.05 (0.21) | 0.46 (0.97)
  Week 12: End of Test (n= 22, 25) | 2.27 (1.59) | 2.92 (1.95)
  Week 12: 2 minutes after end of test (n= 22, 23) | 0.35 (0.68) | 0.65 (1.06)
  Week 16: Resting (n= 19, 23) | 0.13 (0.33) | 0.50 (1.23)
  Week 16: End of Test (n= 18, 23) | 2.50 (1.91) | 2.83 (1.69)
  Week 16: 2 minutes after end of test (n= 19, 23) | 0.41 (0.72) | 0.70 (1.25)
  Week 20: Resting (n= 19, 21) | 0.05 (0.16) | 0.67 (1.14)
  Week 20: End of Test (n= 18,22) | 2.31 (1.70) | 3.11 (2.17)
  Week 20: 2 minutes after end of test (n= 18, 20) | 0.31 (0.55) | 0.75 (1.15)
  Week 24: Resting (n= 20, 21) | 0.18 (0.49) | 0.40 (0.82)
  Week 24: End of Test (n= 20, 21) | 2.58 (1.87) | 2.93 (1.90)
  Week 24: 2 minutes after end of test (n= 20, 20) | 0.29 (0.62) | 0.67 (1.07)

12. Secondary Outcome: Mean Pulmonary Artery Pressure (PAP) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including right Pulmonary Arterial Pressure (PAP). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline breathing ambient air (n=27,28) | 61.7 (15.6) | 59.2 (11.6)
  Baseline every 2 mins breathing NO (1st) (n=20,20) | 61.6 (18.7) | 55.7 (12.0)
  Baseline every 2 mins breathing NO (2nd) (n=17,18) | 58.1 (16.7) | 53.3 (11.5)
  Baseline 5 mins after NO administration (n=20,14) | 60.9 (16.2) | 56.9 (10.8)
  Baseline 15 mins after NO administration(n=19,19) | 60.3 (16.0) | 56.5 (10.3)
  Week 24 breathing ambient air (n=20,22) | 52.5 (11.4) | 55.5 (11.6)
  Week 24 every 2 mins breathing NO (1st) (n=10,13) | 50.9 (17.5) | 55.1 (13.9)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 46.2 (18.1) | 53.9 (14.1)
  Week 24 5 mins after NO administration (n=10,12) | 47.0 (15.8) | 57.5 (12.8)
  Week 24 15 mins after NO administration (n=10,14) | 48.1 (13.7) | 57.2 (12.4)

13. Secondary Outcome: Mean Pulmonary Artery Wedge Pressure (PAWP) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Pulmonary Arterial Wedge Pressure (PAWP). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline breathing ambient air (n=26,28) | 9.0 (2.6) | 7.6 (2.3)
  Baseline every 2 mins breathing NO (1st) (n=20,17) | 9.5 (2.0) | 7.7 (2.9)
  Baseline every 2 mins breathing NO (2nd) (n=17,16) | 9.4 (2.2) | 7.8 (3.4)
  Baseline 5 mins after NO administration (n=19,12) | 9.5 (2.7) | 7.8 (2.9)
  Baseline 15 mins after NO administration(n=18,17) | 9.6 (2.4) | 8.1 (2.6)
  Week 24 breathing ambient air (n=19,22) | 8.4 (3.2) | 8.6 (2.8)
  Week 24 every 2 mins breathing NO (1st) (n=9,13) | 7.9 (3.1) | 10.2 (3.7)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 7.0 (3.4) | 10.0 (3.7)
  Week 24 5 mins after NO administration (n=10,12) | 7.1 (3.1) | 10.3 (3.3)
  Week 24 15 mins after NO administration (n=10,14) | 6.7 (2.8) | 10.4 (3.6)

14. Secondary Outcome: Mean Systolic Arterial Pressure (SAP) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Systolic Arterial Pressure (SAP). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline breathing ambient air (n=26,28) | 110.3 (19.5) | 108.2 (15.4)
  Baseline every 2 mins breathing NO (1st) (n=20,19) | 108.3 (18.9) | 106.9 (18.0)
  Baseline every 2 mins breathing NO (2nd) (n=17,17) | 109.9 (19.1) | 105.4 (18.1)
  Baseline 5 mins after NO administration (n=21,15) | 106.0 (17.7) | 107.1 (18.6)
  Baseline 15 mins after NO administration(n=19,19) | 109.5 (20.3) | 106.9 (16.7)
  Week 24 breathing ambient air (n=20,22) | 108.0 (19.8) | 106.9 (18.8)
  Week 24 every 2 mins breathing NO (1st) (n=10,13) | 103.9 (17.5) | 102.9 (20.4)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 104.8 (18.3) | 103.6 (19.2)
  Week 24 5 mins after NO administration (n=9,12) | 103.4 (18.7) | 104.0 (20.0)
  Week 24 15 mins after NO administration (n=10,14) | 103.8 (21.4) | 107.3 (18.3)

15. Secondary Outcome: Mean Heart Rate (HR) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Heart Rate (HR). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
beats per minute (bpm)
  Baseline breathing ambient air (n=27,28) | 77.3 (7.5) | 84.9 (13.0)
  Baseline every 2 mins breathing NO (1st) (n=20,19) | 75.9 (12.9) | 84.4 (15.5)
  Baseline every 2 mins breathing NO (2nd) (n=17,17) | 75.2 (13.6) | 83.3 (13.2)
  Baseline 5 mins after NO administration (n=19,15) | 73.2 (10.2) | 84.3 (13.9)
  Baseline 15 mins after NO administration(n=18,19) | 76.2 (9.0) | 85.1 (13.8)
  Week 24 breathing ambient air (n=20,22) | 76.6 (8.6) | 83.0 (12.8)
  Week 24 every 2 mins breathing NO (1st) (n=9,13) | 76.3 (10.1) | 82.5 (15.3)
  Week 24 every 2 mins breathing NO (2nd) (n=8,11) | 76.6 (10.3) | 82.8 (16.7)
  Week 24 5 mins after NO administration (n=9,12) | 75.7 (10.2) | 79.3 (10.4)
  Week 24 15 mins after NO administration (n=10,14) | 73.2 (8.3) | 82.9 (10.5)

16. Secondary Outcome: Mean Cardiac Output (CO) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Cardiac Output (CO). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
L/min
  Baseline breathing ambient air (n=27,28) | 4.20 (1.33) | 4.09 (1.44)
  Baseline every 2 mins breathing NO (1st) (n=19,20) | 4.02 (1.32) | 4.22 (1.64)
  Baseline every 2 mins breathing NO (2nd) (n=17,18) | 3.98 (1.16) | 4.43 (1.80)
  Baseline 5 mins after NO administration (n=19,14) | 4.20 (1.16) | 4.71 (1.95)
  Baseline 15 mins after NO administration(n=18,19) | 3.87 (1.03) | 4.47 (2.15)
  Week 24 breathing ambient air (n=20,22) | 4.90 (1.21) | 4.35 (1.57)
  Week 24 every 2 mins breathing NO (1st) (n=10,13) | 4.80 (1.26) | 4.67 (2.27)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 4.79 (1.31) | 4.62 (2.26)
  Week 24 5 mins after NO administration (n=10,12) | 4.63 (1.21) | 4.65 (1.99)
  Week 24 15 mins after NO administration (n=10,14) | 4.48 (1.21) | 4.46 (1.98)

17. Secondary Outcome: Mean Pulmonary Vascular Resistance (PVR) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Pulmonary Vascular Resistance (PVR). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration. PVR calculated according to the equation:PVR = (PAP - PCWP)/CO
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: dyn*s/cm^5
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
dyn*s/cm^5
  Baseline breathing ambient air (n=27,27) | 1124.4 (460.0) | 1118.3 (486.7)
  Baseline every 2 mins breathing NO (1st) (n=19,17) | 1180.9 (520.8) | 1067.9 (509.1)
  Baseline every 2 mins breathing NO (2nd) (n=17,16) | 1064.6 (458.9) | 982.8 (483.9)
  Baseline 5 mins after NO administration (n=19,11) | 1131.5 (491.2) | 1160.4 (510.0)
  Baseline 15 mins after NO administration(n=18,16) | 1181.9 (498.7) | 1132.9 (461.0)
  Week 24 breathing ambient air (n=19,21) | 729.9 (230.1) | 1017.0 (369.1)
  Week 24 every 2 mins breathing NO (1st) (n=9,14) | 706.9 (285.5) | 1000.6 (501.5)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 687.4 (276.3) | 1033.6 (546.2)
  Week 24 5 mins after NO administration (n=10,12) | 717.2 (271.6) | 987.8 (370.4)
  Week 24 15 mins after NO administration (n=10,14) | 776.1 (286.8) | 1042.5 (388.4)

18. Secondary Outcome: Mean Systemic Vascular Resistance (SVR) at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess several prognostic hemodynamic variables in pulmonary hypertension, including Systemic Vascular Resistance (SVR). Were assessed when the patient was in a stable hemodynamic rest state (as demonstrated by three consecutive Mean PAP and CO measurements within 10% of each other). PAP was assessed when the patient was breathing ambient air, every 2 minutes whilst breathing Nitric Oxide(NO) (1st and 2nd), 5 min after the end of NO administration, and 15 mins after the end of NO administration. SVR was calculated according to the equation: SVR = (Paorta - Pright atrium)/CO
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: dyn*s/cm^5
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
dyn*s/cm^5
  Baseline breathing ambient air (n=26,26) | 1674.4 (761.2) | 1764.8 (481.9)
  Baseline every 2 mins breathing NO (1st) (n=18,15) | 1778.2 (709.5) | 1769.7 (457.0)
  Baseline every 2 mins breathing NO (2nd) (n=16,14) | 1807.3 (615.1) | 1664.7 (472.0)
  Baseline 5 mins after NO administration (n=18,11) | 1609.2 (593.4) | 1666.6 (488.6)
  Baseline 15 mins after NO administration(n=17,15) | 1976.3 (877.5) | 1748.4 (499.3)
  Week 24 breathing ambient air (n=18,21) | 1427.2 (446.8) | 1667.9 (357.8)
  Week 24 every 2 mins breathing NO (1st) (n=9,13) | 1344.2 (474.8) | 1579.3 (386.8)
  Week 24 every 2 mins breathing NO (2nd) (n=9,11) | 1367.9 (601.7) | 1592.5 (389.0)
  Week 24 5 mins after NO administration (n=9,12) | 1419.7 (566.6) | 1503.9 (305.3)
  Week 24 15 mins after NO administration (n=10,14) | 1431.7 (524.4) | 1629.3 (355.6)

19. Secondary Outcome: Blood Gas Measurement - PaO2 at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including PaO2 levels at baseline and Study completion Week 24.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline n=22,21 | 63.36 (14.33) | 63.75 (12.02)
  Week 24 n=16,17 | 72.49 (14.09) | 70.13 (16.72)

20. Secondary Outcome: Blood Gas Measurement - PaCO2 at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including PaCO2 levels at baseline and Study completion Week 24.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline n=23,21 | 32.70 (4.40) | 30.02 (4.76)
  Week 24 n=16,17 | 33.36 (5.11) | 30.23 (3.55)

21. Secondary Outcome: Blood Gas Measurement - PvO2 at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including PvO2 levels at baseline and Study completion Week 24.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
mmHg
  Baseline n=14,14 | 33.16 (4.62) | 34.70 (4.75)
  Week 24 n=11,11 | 35.56 (3.80) | 32.65 (4.18)

22. Secondary Outcome: Blood Gas Measurement - Arterial Saturation at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including Arterial Saturation levels at baseline and Study completion Week 24.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
percentage of saturation
  Baseline n=19,16 | 87.99 (9.19) | 91.81 (4.05)
  Week 24 n=14,15 | 92.89 (4.50) | 91.78 (3.36)

23. Secondary Outcome: Blood Gas Measurement - Venous Saturation at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including Venous Saturation levels at baseline and Study completion Week 24.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
percentage of saturation
  Baseline n=17,14 | 57.96 (10.48) | 60.84 (6.61)
  Week 24 n=13,13 | 65.11 (6.91) | 57.00 (9.18)

24. Secondary Outcome: Blood Gas Measurement - pH at Baseline and Study Completion
Description: The right heart catheter assessment was performed to assess Blood Gas Measurements in pulmonary hypertension, including pH levels at baseline and Study completion Week 24. The pH scale measures how acidic or basic a substance is. It ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic.
Time Frame: Baseline, and Study completion (Week 24)
Population: The intention to treat population (ITT) will include all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: pH scale
Arm/Group | STI571 | Placebo
Number analyzed (Participants) | 28 | 31
pH scale
  Baseline n=24,23 | 7.43 (0.04) | 7.44 (0.05)
  Week 24 n=17,17 | 7.44 (0.05) | 7.46 (0.05)

ADVERSE EVENTS:
Groups:
- Core - STI571: Core - STI571
- Core - Placebo: Core - Placebo
- Extension - STI571: Extension - STI571
Arm/Group | Core - STI571 | Core - Placebo | Extension - STI571
Serious Adverse Events (participants affected / at risk) | 12/28 | 11/31 | 16/22
Other Adverse Events (participants affected / at risk) | 26/28 | 25/31 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core - STI571 (N=28) | Core - Placebo (N=31) | Extension - STI571 (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 0 | 1
Catheter related complication (General disorders) | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 7
General physical health deterioration (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 1 | 1
Syncope (Nervous system disorders) | 2 | 1 | 3
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 0 | 1
Arterial rupture (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core - STI571 (N=28) | Core - Placebo (N=31) | Extension - STI571 (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 0 | 2
Palpitations (Cardiac disorders) | 3 | 4 | 4
Pericardial effusion (Cardiac disorders) | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 4 | 4 | 8
Hypothyroidism (Endocrine disorders) | 0 | 0 | 4
Eye swelling (Eye disorders) | 3 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 4
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 14 | 5 | 8
Vomiting (Gastrointestinal disorders) | 6 | 1 | 3
Asthenia (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 2 | 3 | 4
Chest pain (General disorders) | 1 | 3 | 1
Exercise tolerance decreased (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 3 | 4 | 3
General physical health deterioration (General disorders) | 1 | 0 | 3
Oedema (General disorders) | 1 | 0 | 8
Oedema peripheral (General disorders) | 7 | 5 | 9
Pain (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 4
Bacteriuria (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2
Cystitis (Infections and infestations) | 0 | 1 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 5
Helicobacter infection (Infections and infestations) | 0 | 0 | 2
Herpes simplex (Infections and infestations) | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 8 | 14
Oral candidiasis (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 6 | 1 | 11
Sinusitis (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0
Blood amylase increased (Investigations) | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 3
Blood creatinine increased (Investigations) | 1 | 0 | 3
Blood potassium decreased (Investigations) | 3 | 0 | 6
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 3
C-reactive protein increased (Investigations) | 0 | 1 | 3
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 2 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Dizziness (Nervous system disorders) | 3 | 3 | 5
Headache (Nervous system disorders) | 10 | 6 | 4
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0 | 4
Sleep disorder (Psychiatric disorders) | 2 | 0 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Flushing (Vascular disorders) | 2 | 3 | 0
Haematoma (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.